CLINICAL TRIAL: NCT06366230
Title: Adding Urea to the Final Dialysis Fluid in Order to Prevent Dialysis Disequilibrium in Patients Who Need Aggressive Dialysis for Electrolyte Abnormalities
Brief Title: Adding Urea to the Final Dialysis Fluid
Acronym: Urea dialysate
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-41450
Record Dates: First submitted 2024-04-04; First posted 2024-04-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Dysequilibrium Syndrome; ESRD; Hyperkalemia; Metabolic Acidosis
Keywords: ESRD; Urea; Disequilibrium; Potassium; Acid/base
MeSH Terms: conditions — Dysequilibrium syndrome; Kidney Failure, Chronic; Hyperkalemia; Acidosis | interventions — Urea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Urea dialysate (Experimental): Patients who had urea added to the final dialysis fluid
  Interventions: Drug: Urea in the dialysate

INTERVENTIONS:
Drug: Urea in the dialysate — Adding urea to the dialysis fluid. Ure-Na 15 grams would be used. It would be added to the acid component of the dialysis fluid. The amount added would depend on the serum BUN concentration and is determined by a simple calculation. It would be available in powder form. Urea would be added just to the first 1-3 dialysis treatments as needed.
  Other Names: Ure-Na

SUMMARY:
At times patients with advanced renal failure present with severe hyperkalemia or acidosis and very high serum blood urea nitrogen (BUN) concentrations. These patients cannot be dialyzed aggressively as the lowering of serum BUN may results in disequilibrium syndrome but on the other hand they need aggressive dialysis in order to lower their serum potassium or fix their severe acidosis. If one is able to add urea to the dialysis fluid, one can prevent the rapid lowering of serum BUN and osmolality at the same time as doing aggressive dialysis to lower serum potassium and/or fix the metabolic acidosis.

DETAILED DESCRIPTION:
Ure-Na 15 gram tablets would be used to add to the dialysis fluid How much urea to add would be a simple calculation based on the 45X dialysis system and the patients serum urea concentration. The dialysate fluid urea concentration would be made to be about 15-40 mg/dL lower than the serum concentration. The patients labs/vitals and symptoms would be closely monitored throughout the dialysis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Serum Urea > 120
* Serum Potassium > 5.5 or serum CO2 < 15 or need for aggressive dialysis due to toxic ingestion
* need for dialysis

Exclusion Criteria:

* Pediatric
* need for CRRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Disequilibrium | within 24 hours after starting dialysis
  Dialysis disequilibrium syndrome (DDS) refers to an array of neurological manifestations that are seen during or following dialysis. The symptoms can range from headache, nausea, blurred vision, restlessness and confusion to coma and seizures in rare cases. The physician will assess DDS.
Serum potassium concentration | Potassium levels every 6 hours for 24 hours after end of dialysis
  Improvement in serum potassium concentration in mEq/L would be measured and documented with the study
Serum CO2 concentration | Serum CO2 levels every 6 hours for 24 hours after end of dialysis
  Improvement in metabolic acidosis would be monitored by checking serum CO2 concentration in mEq/L

SECONDARY OUTCOMES:
Serum BUN concentration | Serum BUN concentration twice a day for 3 days
  The trend in serum BUN concentration in mg/dL would be followed

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Sam, MD, Principal Investigator — Zuckerberg San Francisco General- UCSF
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No